CLINICAL TRIAL: NCT04476602
Title: Ambulatory Management of Moderate to High Risk COVID-19 (SARS-CoV-2) Patients - The Coronavirus Related Outpatient Work Navigators (CROWN) Protocol
Acronym: CROWN
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Gita Lisker, Physician, Northwell Health
Other Study IDs: 20-0618
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Covid-19 (SARS-CoV-2)
Keywords: COVID-19 (SARS-CoV-2); Homecare; Ambulatory
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 (SARS-CoV-2) patients: adults 18 or older, ambulatory , with COVID-19 (SARS-CoV-2)

SUMMARY:
Descriptive report of the Northwell CROWN program for ambulatory treatment of COVID-19 (SARS-CoV-2) patients with moderate to high risk features

DETAILED DESCRIPTION:
At the peak of the COVID-19 (SARS-CoV-2) pandemic in New York City, there was a shortage of hospital resources as well as a fear among many New Yorkers of going to the hospital. Emergency Services dead on arrival calls increased by as much as eight-fold.We created the CROWN Program, a pulmonary physician guided home-care protocol to treat ambulatory COVID-19 (SARS-CoV-2) patients with moderate to high risk features. This is a retrospective review of our CROWN program's patient characteristics, results and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 (SARS-CoV-2) infection Ambulatory

Exclusion Criteria:

* Need for hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General public
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Hospital Admission | 30 days
  admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Gita Lisker, MD, Principal Investigator — Northwell Health; ramona ramdeo, Study Director — Northwell Health
Locations (1):
- 410 Lakeville Road, Suite 107, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No